CLINICAL TRIAL: NCT01531140
Title: High-volume Polyethylene Glycol Solution (PEG) Versus Low-volume PEG Plus Stimulant Laxative Versus Sennosides for Colon Cleansing Before Colonoscopy: a Randomized, Single Blinded Study
Brief Title: PEG Versus PEG+Bisacodyl Versus Sennosides for Colon Cleansing Before Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2012
Record Dates: First submitted 2012-01-16; First posted 2012-02-10 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-01

CONDITIONS: Colonoscopy Preparation
Keywords: colonoscopy cleansing; PEG; sennosides; children
MeSH Terms: interventions — Polyethylene Glycols; Sennosides

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Polyethylene glycol (Active Comparator): Polyethylene glycol p.o.(Fortrans):60 ml/kg for 2 days
  Interventions: Drug: Polyethylene glycol
- PEG + Bisacodyl (Experimental): Polyethylene glycol p.o.(Fortrans): 30 ml/kg for 2 days + Bisacodyl p.o.: 10-15 mg/day
  Interventions: Drug: polyethylene glycol +Bisacodyl
- Sennosides (Experimental): Sennosides: 1tbl/8kg/day for 2 days (1 tbl=8,6 mg sennosides B)
  Interventions: Drug: Sennosides

INTERVENTIONS:
Drug: polyethylene glycol +Bisacodyl — Polyethylene glycol (Fortrans) p.o. 30 ml/kg/2days + Bisacodyl p.o.10-15 mg/day for 2 days
  Other Names: Polyethylene glycol: Fortrans
  Arms: PEG + Bisacodyl
Drug: Polyethylene glycol — Polyethylene glycol p.o.: 60 ml/kg/days
  Other Names: Polyethylene glycol: Fortrans
  Arms: Polyethylene glycol
Drug: Sennosides — Sennosides 1tbl/8kg for 2 days
  Other Names: Sennosides: Xenna
  Arms: Sennosides

SUMMARY:
Background:

Polyethylene glycol (PEG) solution has been proven to be effective for large bowel cleansing prior to colonoscopy in children. However, the high volume of fluid and its taste sometimes lead to inappropriate cleansing of the bowel, thus search for other bowel preparation is needed.

Aim:

The efficacy and tolerability of three different bowel cleansing protocols used in children for colonoscopy: high-volume PEG compared with low-volume PEG with stimulant laxative (bisacodyl) compared with sennosides.

Methods:

Participants aged 10-18 years will be randomly assigned to receive either PEG 60 ml/kg/day or PEG 30 ml/kg/day plus oral bisacodyl 10-15 mg/day or sennosides 2mg/kg/day for 2 days prior to the colonoscopy. The outcome measures will be:bowel cleansing efficacy, scored by a blinded endoscopist using the Ottawa scale and Aronchick Scale (the mean total score, proportions of participants with excellent/good and with poor/inadequate bowel preparation), and the patient satisfaction score(0-10)with the method of preparation for the colonoscopy evaluated with the visual analog scale. Analysis will be done on an intention to treat basis.

DETAILED DESCRIPTION:
Patients are excluded if they had known allergy to one of the tested preparations such as bisacodyl (Bisacodyl VP, ICN Polfa, Rzeszow, Poland), polyethylene glycol (Fortrans, Beaufour Ipsen Industry, Dreux, France) and/or sennoside (Xenna Extra, US Pharmacia, Wroclaw, Poland) and had disorders that make oral intake of the preparation impossible (neurological disorders, intestinal obstruction, mental retardation etc.).

Study design:

On admission day patients are allocated to one of the groups by study investigators, according to the randomization list created by an independent person using block randomization by a standard statistical program StatsDirect [version 2,3,8 (2005)] (6 patients were included in each block).

During the preparation for colonoscopy each patient are observed for procedure tolerance. On the day of endoscopy, each patient evaluated the degree of the acceptance of the method of bowel cleaning (according to visual analog scale (VAS) and the occurrence of side effects (diary). The endoscopist performing colonoscopy, blinded for the bowel preparation regimen evaluate bowel cleansing and score it, according to the Aronchick and Ottawa scale. The rate of cecum intubation, and the colonoscopy complications (defined as bowel perforation and/or significant bleeding) are analyzed in each bowel preparation group.

ELIGIBILITY:
Inclusion Criteria:

* children 10 - 18 years of age referred for colonoscopy
* informed consent signed

Exclusion Criteria:

* allergy to PEG, sennosides or bisacodyl
* disorders that make oral intake of the preparation impossible (neurological disorders, intestinal obstruction, mental retardation etc.)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 240 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
proportions of participants with good or excellent bowel preparation assessed with Ottawa Scale | bowel preparation quality with Ottawa scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to the Ottawa scale the quality of bowel preparation is estimated by adding points for the cleansing of three parts of colon (descending, transversal and ascending) and points for amount of fluid in the bowel. Score: 0-1 - excellent cleansing, 2-4 - good, 5-7 - sufficient, 8-10 - poor, 11-14 - not appropriate.
proportions of participants with poor/inadequate bowel preparation assessed with Ottawa Scale | bowel preparation quality with Ottawa scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to the Ottawa scale the quality of bowel preparation is estimated by adding points for the cleansing of three parts of colon (descending, transversal and ascending) and points for amount of fluid in the bowel. Score: 0-1 - excellent cleansing, 2-4 - good, 5-7 - sufficient, 8-10 - poor, 11-14 - not appropriate.

SECONDARY OUTCOMES:
proportions of participants with very good/good bowel preparation assessed with Aronchick Scale | bowel preparation quality with Aronchick scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to Aronchick scale preparation is estimated as:
  * very good: small amount of clear fluid is present, more than 95% mucosa is visible
  * good: small amount of clear fluid easy to suction away or flush is present, more than 90% of mucosa is visible
  * sufficient: big amount of clear fluid covering 5-25% of mucosa, more than 90% of mucosa visible
  * poor: semi-liquid stool that cannot be flushed, less than 90% of mucosa visible
  * inadequate: colonoscopy must be repeated
proportions of participants with poor/inadequate bowel preparation assessed with Aronchick Scale | bowel preparation quality with Aronchick scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to Aronchick scale preparation is estimated as:
  * very good: small amount of clear fluid is present, more than 95% mucosa is visible
  * good: small amount of clear fluid easy to suction away or flush is present, more than 90% of mucosa is visible
  * sufficient: big amount of clear fluid covering 5-25% of mucosa, more than 90% of mucosa visible
  * poor: semi-liquid stool that cannot be flushed, less than 90% of mucosa visible
  * inadequate: colonoscopy must be repeated
mean bowel preparation score assessed with Ottawa Scale | bowel preparation quality with Ottawa scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to the Ottawa scale the quality of bowel preparation is estimated by adding points for the cleansing of three parts of colon (descending, transversal and ascending) and points for amount of fluid in the bowel. Score: 0-1 - excellent cleansing, 2-4 - good, 5-7 - sufficient, 8-10 - poor, 11-14 - not appropriate.
mean bowel preparation score assessed with Aronchick scale | bowel preparation quality with Aronchick scale is assesed during colonoscopy (3rd day of the study) by endoscopist blinded for the method of preparation
  According to Aronchick scale preparation is estimated as:
  * very good: small amount of clear fluid is present, more than 95% mucosa is visible
  * good: small amount of clear fluid easy to suction away or flush is present, more than 90% of mucosa is visible
  * sufficient: big amount of clear fluid covering 5-25% of mucosa, more than 90% of mucosa visible
  * poor: semi-liquid stool that cannot be flushed, less than 90% of mucosa visible
  * inadequate: colonoscopy must be repeated
patient satisfaction with the method of preparation assessed with Visual analogue scale (VAS) | assessed by patient after completion of bowel preparation regimen before colonoscopy (3rd day of the study)
  VAS scale is horizontal line 100 mm lenght anchored by word description at each end (very good, very bad).The patient mark on the line the point that feel represent the perception of bowel preparation regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Dziechciarz, MD, Study Chair — Medical University of Warsaw; Jaroslaw Kierkus, MD, Principal Investigator — Child Health Center
Locations (2):
- Poland (2):
  - Warsaw Medical University, Warsaw
  - Child Health Center, Warsaw